CLINICAL TRIAL: NCT00969254
Title: Phase III Clinical Study, Prospective, Multicenter, Double-blind, Randomized, Double-dummy to Assess the Efficacy and Safety of "Pílulas de Lussen®" Compared to the Pyridium® in the Symptomatic Control of Dysuria
Brief Title: Study to Assess the Efficacy and Safety of "Pílulas de Lussen®" Compared to the Pyridium® in the Symptomatic Control of Dysuria
Acronym: E01OSMPLS0108
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratorios Osorio de Moraes Ltda. (Industry)
Responsible Party: Maria Angelina Nardy Mattos, Laboratórios Osório de Moraes Ltda.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E01-OSM-PLS-01-08
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Dysuria
Keywords: Pílulas de Lussen; Efficacy; Safety; Dysuria; Symptomatic control
MeSH Terms: conditions — Dysuria | interventions — Phenazopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pílulas de Lussen (Experimental): Take one dragee of drug A* and one dragee of drug B** every 8 hours for three days.
  * Drug A: Pílulas de Lussen®
  ** Drug B: placebo.
  Interventions: Drug: Pílulas de Lussen
- Pyridium® (Active Comparator): Take one dragee of drug A* and one dragee of drug B** every 8 hours for three days.
  * Drug A: Pyridium®
  ** Drug B: placebo.
  Interventions: Drug: Pyridium®

INTERVENTIONS:
Drug: Pílulas de Lussen — Take one dragee of drug A* and one dragee of drug B** every 8 hours for three days.
  * Drug A: Pílulas de Lussen®
  ** Drug B: placebo.
  Arms: Pílulas de Lussen
Drug: Pyridium® — Take one dragee of drug A* and one dragee of drug B** every 8 hours for three days.
  * Drug A: Pyridium®
  ** Drug B: placebo.
  Arms: Pyridium®

SUMMARY:
Clinical Study, prospective, comparative, randomized, double-dummy entry with random from a total of 80 patients, 40 patients will receive the test medication (Pílulas de Lussen®) plus placebo and 40 patients will receive the comparative (Pyridium®) plus placebo.

DETAILED DESCRIPTION:
Phase III Clinical Study, prospective, multicenter, double-blind, randomized, double-dummy to assess the efficacy and safety of "Pílulas de Lussen®" compared to the Pyridium® in the symptomatic control of dysuria in 80 patients of either sex or race, older than 18 years, with symptoms of dysuria, 40 patients will receive the test medication (Pílulas de Lussen®) plus placebo and 40 patients will receive the comparative (Pyridium®) plus placebo to evaluate the effectiveness and tolerability of 'Pílulas de Lussen' for symptomatic relief of dysuria.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years;
* Patients with symptoms of dysuria characterized by pain/burning sensation in the lower urinary tract and discomfort in urination;
* Patients who are female and are of childbearing age should use reliable method of contraception and have negative pregnancy test.
* Patients who consent to participate in the study.

Exclusion Criteria:

* Patients with sensitivity to any component of the formula;
* Patients pregnant or lactating;
* Patients with a history of glaucoma, heart failure, cardiac arrhythmias, prostatic hypertrophy, paralytic ileus or pyloric stenosis;
* Patients with menorrhagia or heavy menstrual periods;
* Patients who need to use antibiotics or chemotherapy;
* Patients who can not follow the procedures shown in this Clinical Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogic Scale and opinion of the investigator. | 3 days

SECONDARY OUTCOMES:
Of adverse events related to study medication by the Naranjo Algorithm. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Lúcia Hime, Principal Investigator — Universidade de Santo Amaro (UNISA); Nabil Ghorayeb, Principal Investigator — Clínica Nabil Ghorayeb; Patrícia Smith, Principal Investigator — Clínica Nabil Ghorayeb; Ceci Lopes, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HCFMUSP)